CLINICAL TRIAL: NCT03009487
Title: A Multi-center, Randomized, Double-blind, Phase III Clinical Trial to Evaluate the Efficacy and Safety of Olmesartan/Amlodipine/Rosuvastatin Combination Treatment in Patients With Concomitant Hypertension and Hyperlipidemia
Brief Title: A Clinical Trial to Evaluate the Efficacy and Safety of Olmesartan/Amlodipine/Rosuvastatin Combination Treatment in Patients With Concomitant Hypertension and Hyperlipidemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DW_DWJ1351003
Record Dates: First submitted 2016-12-12; First posted 2017-01-04 (Estimated); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Hypertension; Hyperlipidemias
MeSH Terms: conditions — Hypertension; Hyperlipidemias | interventions — Amlodipine; olmesartan; Drug Combinations; Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Amlodpine, Olmesartan, Rosuvastatin (Experimental): co-administration of Olmesartan, Amlodipine and Rosuvastatin
  Interventions: Drug: Amlodipine/Olmesartan 10/40mg (Combination drug), Rosuvastatin 20mg
- Olmesartan, Rosuvastatin (Placebo Comparator): co-administration of Olmesartan and Rosuvastatin
  Interventions: Drug: Olmesartan 40 mg, Rosuvastatin 20mg
- Amlodipine, Olmesartan (Placebo Comparator): co-administration of Amlodipine and and Olmesartan
  Interventions: Drug: Amlodipine/Olmesartan 10/40mg (Combination drug)

INTERVENTIONS:
Drug: Amlodipine/Olmesartan 10/40mg (Combination drug), Rosuvastatin 20mg — co-administration of Sevikar tab. 10/40mg(Amlodipine/Olmesartan 10/40mg), Crestor Tab. 20mg(Rosuvastatin 20mg) and placebo of Olmesartan 40mg
  Arms: Amlodpine, Olmesartan, Rosuvastatin
Drug: Olmesartan 40 mg, Rosuvastatin 20mg — co-administration of Olmetec tab. 40mg(Olmesartan 40mg), Crestor tab. 20mg(Rosuvastatin 20mg) and placebo of Sevikar Tab 10/40mg(Amlodipine/Olmesartan 10/40mg).
  Arms: Olmesartan, Rosuvastatin
Drug: Amlodipine/Olmesartan 10/40mg (Combination drug) — co-administration of Sevikar tab. 10/40mg(Amlodipine/Olmesartan 10/40mg) 10/40mg, Placebo of Olmesartan Tab. 40mg and Placebo of Rosuvastatin 20mg
  Arms: Amlodipine, Olmesartan

SUMMARY:
A multi-center, randomized, double-blind, phase III clinical trial to evaluate the efficacy and safety of Olmesartan/Amlodipine/Rosuvastatin combination treatment in patients with concomitant hypertension and hyperlipidemia

ELIGIBILITY:
Inclusion Criteria:

* Age 20 to 80 years
* patients with hypertension and hyperlipidemias

Exclusion Criteria:

* orthostatic hypotension
* History of ventricular tachycardia, atrial fibrillation
* uncontrolled diabetes mellitus

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 265 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
the change of sitSBP based on baseline between Treatment arm and control 1 arm | 8 weeks
the change of LDL-C based on baseline between Treatment arm and control2 arm | 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul national university bundang hospital, Seoul, South Korea